CLINICAL TRIAL: NCT00270972
Title: A Confirmatory Study to Evaluate the Safety and Efficacy of Cryopreserved Bilayered Cellular Matrix (ORCEL) for the Treatment of Venous Ulcers
Brief Title: The Evaluation of OrCel for the Treatment of Venous Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ortec International (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-VLU-02-CLN
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2006-06-05 (Estimated); Status verified 2006-06

CONDITIONS: Venous Insufficiency; Leg Ulcer
Keywords: Venous leg ulcer; Venous insufficiency; OrCel
MeSH Terms: conditions — Venous Insufficiency; Leg Ulcer; Varicose Ulcer

INTERVENTIONS:
Device: Bilayered Cellular Matrix (OrCel)

SUMMARY:
This study was designed to confirm the clinical benefits and safety of OrCel in the treatment of venous ulcers. OrCel and standard care are compared to standard care alone. Standard care consists of currently accepted compression therapy.

Patients are treated for 12 weeks. Patients with healed ulcers are followed for an additional 12 weeks to assess durability of the healed wound.

ELIGIBILITY:
Inclusion Criteria:

* Any race, between 18 and 85 years of age
* Male or female
* Chronic venous insufficiency
* Ulcer size between 2 and 20 sq cm, inclusive
* Ulcer present for at least one month
* ABI >0.7

Exclusion Criteria:

* Decrease in wound size >35% during Screening Phase
* Infection at ulcer site
* Uncontrolled diabetes mellitus
* Malnutrition
* Previous treatment with excluded medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-09

PRIMARY OUTCOMES:
Investigator Assessment of wound healing

SECONDARY OUTCOMES:
Planimetric assessment of wound healing
Photographic assessment of wound healing

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Baptist Medical Center South, Montgomery, Alabama
  - Associated Foot and Ankle Specialists, Phoenix, Arizona
  - Eden Podiatry Group, Castro Valley, California
  - PPH Center for Wound Care and Hyperbaric Medicine, Poway, California
  - Wound Healing Center, Terre Haute, Indiana
  - Southside Hospital, Bay Shore, New York
  - St Luke's Roosevelt, New York, New York
  - Center for Advanced Wound Care, Reading, Pennsylvania
  - Warren General Hospital, Warren, Pennsylvania
  - Hyperbaric and Wound Care Associates, Milwaukee, Wisconsin